CLINICAL TRIAL: NCT00751790
Title: A Multicenter, Open, Non-comparative, Phase III Study on the Efficacy, Pharmacokinetics and Safety of Two Injections of Triptorelin Embonate 22.5 mg 6-month Formulation in Patients With Advanced Prostate Cancer.
Brief Title: Efficacy and Safety of a Triptorelin 6-month Formulation in Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEB-TRI6M-301
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Results first posted 2012-06-13 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2012-08

CONDITIONS: Prostatic Neoplasm
Keywords: triptorelin, 6-month formulation, advanced prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triptorelin (Experimental)
  Interventions: Drug: triptorelin embonate (INN)

INTERVENTIONS:
Drug: triptorelin embonate (INN) — Triptorelin embonate 22.5 mg 6 month formulation to be injected every 24 weeks

SUMMARY:
Efficacy and safety of a triptorelin 6-month formulation in patients with advanced prostate cancer. It was assumed that during the study treatment >90% of the patients would achieve and maintain castrate levels of serum testosterone.

DETAILED DESCRIPTION:
Efficacy of triptorelin treatment on gonadotropin (LH) stimulation from hypophysis, as well as on the PSA (prostate specific antigen) levels and safety laboratory parameters. The triptorelin pharmacokinetics and testosterone pharmacodynamics were assessed in a subset of 15 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven prostate cancer.
* The prostate cancer should be staged T3-4NxMx or TxN1-3Mx or TxNxM1 according to the TNM classification or the patient should have rising PSA after failed local therapy and be candidate for androgen deprivation therapy.
* Serum testosterone levels >5 nmol/L.
* Karnofsky performance index >40.
* Expected survival > 18 months.
* Absence of another malignancy, other than local dermatological, for the previous 5 years.
* Signed informed consent before entry into the study.

Exclusion Criteria:

* Prior hormonal treatment for prostate cancer within 6 months prior to study start.
* Use of finasteride (Proscar®) or dutasteride (Avodart®/Avolve®) within 2 months prior to study start.
* Presence of another neoplastic lesion or brain metastases.
* Prior hypophysectomy or adrenalectomy.
* Known or suspicion of vertebral metastases with risk of spinal compression.
* Severe kidney or liver failure (creatinine > 2 times the upper normal limit, ASAT and ALAT >3 times the upper normal limit).
* Any concomitant disorder or resulting therapy that is likely to interfere with patient compliance or with the study in the opinion of the Investigator.
* Participation in another study with an experimental drug within 3 months before study start or within 5 drug half-lives of the investigational drug (whichever is the longer).
* Known hypersensitivity to any of the test materials or related compounds.
* Known active use of recreational drug or alcohol dependence in the opinion of the Investigator.
* Any current use or use within 6 months prior to treatment start of medications which are known to affect the metabolism and/or secretion of androgenic hormones: ketoconazole, aminoglutethimide, oestrogens, and progesterone.
* Use of systemic or inhaled corticosteroids (topical application permitted).
* Use of anticoagulants: heparin and coumarine derivatives (acetylsalicylic acid permitted).
* Inability to give Informed Consent or to comply fully with the protocol.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles South Africa, Lyttelton Manor, Centurion, South Africa

REFERENCES:
- [Derived] Lundstrom EA, Rencken RK, van Wyk JH, Coetzee LJ, Bahlmann JC, Reif S, Strasheim EA, Bigalke MC, Pontin AR, Goedhals L, Steyn DG, Heyns CF, Aldera LA, Mackenzie TM, Purcea D, Grosgurin PY, Porchet HC. Triptorelin 6-month formulation in the management of patients with locally advanced and metastatic prostate cancer: an open-label, non-comparative, multicentre, phase III study. Clin Drug Investig. 2009;29(12):757-65. doi: 10.2165/11319690-000000000-00000. PMID 19888782

RESULTS

PARTICIPANT FLOW:
Groups:
- Triptorelin: Each subject received 2 injections of Triptorelin 22.5 mg at an interval of 24 weeks
Period: Overall Study
Arm/Group | Triptorelin
Started | 120
Completed | 115
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Triptorelin
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.11 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 120
Region of Enrollment [Number; unit: participants]
  South Africa | 120

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Castration and Maintenance of Castration
Description: Percentage of patients achieving castrate testosterone levels (≤1.735 nmol/L) by Day 29 (28 days after study drug injection) and percentage of patients maintaining castrate testosterone levels from Month 2 to end of Month 12 (Week 48).
Time Frame: at Day 29
Measure: Number; unit: percentage of enrolled patients
Arm/Group | Triptorelin
Number analyzed (Participants) | 120
percentage of enrolled patients | 97.5

2. Secondary Outcome: LH Increase
Description: % of patients showing ≤1.0 IU/L increase in s-LH from 0 to 2 h after 1st & 2nd injection.% changes in PSA throughout treatment.% of 60 pts with s-testosterone levels >1.735 nmol/L after 2nd injection.Testosterone PD and triptorelin PK metrics in 15 pts
Time Frame: day 1 and day 169
Reporting Status: Not Posted
Measure: Number; unit: patient

ADVERSE EVENTS:
Arm/Group | Triptorelin
Serious Adverse Events (participants affected / at risk) | 17/120
Other Adverse Events (participants affected / at risk) | 115/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin (N=120)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Diabetes mellitus (Endocrine disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin (N=120)
Oedema peripheral (General disorders) | 6 (6)
Bronchitis (Infections and infestations) | 6 (7)
Influenza (Infections and infestations) | 19 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (12)
Headache (Nervous system disorders) | 9 (9)
Insomnia (Psychiatric disorders) | 6 (7)
Urinary retention (Renal and urinary disorders) | 6 (10)
Urinary tract infection (Renal and urinary disorders) | 11 (14)
Erectile dysfunction (Reproductive system and breast disorders) | 12 (12)
Testicular atrophy (Reproductive system and breast disorders) | 9 (9)
Hot flush (Vascular disorders) | 87 (98)
Hypertension (Vascular disorders) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or scientific communication related to this study can only take place once the agreement between the Sponsor and the Investigator has been reached.